CLINICAL TRIAL: NCT04597047
Title: A Multicenter Covid-19 Study Conducted to Evaluate the Agreement Between Fingerstick Whole Blood, Venous Whole Blood, Plasma & Serum as Determined on the LumiraDx POC SARS-CoV-2 Ab Test & to Evaluate the Ease of Use at Point of Care Sites
Brief Title: Research & Evaluation of LumiraDx SARS-CoV-2 (COVID-19) Point of Care Ab Test
Acronym: CAPTURE-2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: LumiraDx UK Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S-CLIN-PROT-0031
Record Dates: First submitted 2020-10-19; First posted 2020-10-22 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Covid19
Keywords: POC; SARS-CoV-2; Antibody
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Participants are asked to provide Capillary and Venous Blood Samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- All Patients: (Other): Capillary and Venous Blood Collections
  Interventions: Diagnostic Test: Capillary Collection & Testing; Diagnostic Test: Venous Draw & Testing

INTERVENTIONS:
Diagnostic Test: Capillary Collection & Testing — Two (2) fingersticks will be performed on each subject and capillary blood tested in the LumiraDx SARS-CoV-2 Ab test
Diagnostic Test: Venous Draw & Testing — One (1) Venous Draw (to include one (1) 6.0 mL EDTA tube and one (1) 3.5 mL serum separator tube) will be collected from each subject. Blood will be tested in the LumiraDx SARS-CoV-2 Ab test

SUMMARY:
Evaluation of the agreement between fingerstick samples, venous blood, serum and plasma samples when using the LumiraDx SARS-CoV-2 Ab Test against the reference method, using standard qualitative comparison techniques.

DETAILED DESCRIPTION:
This is a prospective, multi-centre study. One (1) Reference Lab and approximately six (6) Healthcare or Research Facilities within geographic areas experiencing current Covid-19 outbreaks in the U.S. will participate in the study. Study sites may be Point of Care (POC) locations, such as physician office laboratories, urgent care and outpatient clinics, or dedicated research sites.

A subject's participation in this study will consist of a single visit. Following completion of the informed consent process and a review of Inclusion/Exclusion criteria to determine eligibility, each subject will receive a unique study identification number.

Subjects will undergo two (2) fingerstick lancing's and 1 (one) venous blood draw. A total of eleven (11) tests (LumiraDx SARS-CoV-2 Ab and haematocrit) will then be performed using these samples. Specimens will be obtained from each subject enrolled using standard collection methods.

All operators at a site level performing the LumiraDx SARS-CoV-2 Ab POC Test in this study will be required to complete training detailing the running of the LumiraDx Test/Instrument. This will be completed as part of a familiarization period and all operators will be required to show proficiency in using the system for QC, fingerstick, whole blood, plasma and serum testing prior to testing subjects. This will be captured on relevant training forms as part of the site initiation visit. In addition, the operator's satisfaction and ease of use of the LumiraDx SARS-CoV-2 Ab Test will be evaluated by completing an Intended Use Operator Questionnaire.

The LumiraDx SARS-CoV-2 Ab POC Testing will be performed at the site on the same day as the date of collection. Samples will be shipped to a central laboratory for reference testing. Testing in the reference laboratory will be performed by trained laboratory personnel.

Approximately 200 subjects will be enrolled in this study. Approximately thirty (30) SARS-CoV-2 positive, and thirty (30) samples negative for SARS-CoV-2 will be enrolled at each site.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged ≥ 2 years.
2. The subject must have a documented SARS-CoV-2 PCR test in the past 7-30 days. (subjects must be 14+ days post symptom onset at the time of recruitment).
3. Written informed consent must be obtained prior to study enrollment.

   1. A subject who is 18 years or older must be willing to give written informed consent and must agree to comply with study procedures.
   2. The Legal Guardian or Legal Authorized Representative of a subject who is under the age of 18 must give written informed consent and agree to comply with study procedures. Active written assent should be obtained from children of appropriate intellectual age (as defined by the IRB).

Exclusion Criteria:

1. Skin lesions or conditions that would preclude a fingerstick and or a venous blood draw.
2. The subject is currently receiving or has received within the past thirty (30) days of the study visit an experimental biologic, drug, or device including either treatment or therapy.
3. The subject has previously participated in this research study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Performance Evaluation | 4 months
  Evaluation of the agreement between fingerstick samples and venous blood samples on the device; and venous blood, serum and plasma samples on the device versus reference method, using standard qualitative comparison techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Vicki Kalen, Principal Investigator — Eclipse Clinical Research; William Simon, Principal Investigator — Professional Research Network of Kansas; Matthew Morgan, Principal Investigator — Centura Health Physician Group; Melanie Hoppers, Principal Investigator — Physicians Quality Care of Jackson
Locations (4):
- United States (4):
  - Eclipse Clinical Research, Tucson, Arizona
  - Centura Health Physician Group, Northglenn Office, Northglenn, Colorado
  - Professional Research Network of Kansas, Wichita, Kansas
  - Physicians Quality Care of Jackson, Jackson, Tennessee

IPD SHARING:
Plan to Share IPD: No